CLINICAL TRIAL: NCT06409624
Title: Association Between Biomarkers and Kidney Function Decline in Patients With Pulmonary Hypertension
Brief Title: Association Between Biomarkers and Kidney Function Decline in Pulmonary Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: AZ174/18
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Hypertension; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary hypertension: Patients with diagnosed PH by right heart catheterization with or without PH-specific treatment
  Interventions: Other: No intervention is planned as part of the study
- No pulmonary hypertension: Patients in whom PH was excluded by right heart catheterization
  Interventions: Other: No intervention is planned as part of the study

INTERVENTIONS:
Other: No intervention is planned as part of the study — No intervention is planned as part of the study

SUMMARY:
The objective of this study is to examine the association between urinary and plasma biomarkers and change in estimated glomerular filtration rate (eGFR) among patients with pulmonary hypertension (PH).

DETAILED DESCRIPTION:
PH is a severe, progressive disease associated with right ventricular dysfunction, right-sided heart failure (HF) and death. Kidney disease is present in approximately 35% of patients with PH, and its presence is associated with an enhanced risk for adverse outcomes, with the risk increasing incrementally with declining kidney function. Poor right ventricular function may increase venous congestion, alter ventricular interdependence, decrease effective cardiac output and activate the renin-angiotensin- aldosterone system, thereby aggravating kidney disease.

There is a crucial need to better understand the pathophysiological mechanisms linking the failing right heart and the kidney. To date, diagnostic and prognostic biomarkers of kidney disease in PH are lacking. The objective of this study is to examine the association between urinary and plasma biomarkers and change in eGFR among patients with PH.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients aged ≥18 years
* Undergoing right heart catheterization (RHC)

Exclusion Criteria:

* Active tumor disease requiring targeted therapy
* inflammatory or autoimmune disease with renal involvement requiring systemic immunosuppressive treatment
* unexplained kidney function decline, defined as serum creatinine increase ≥0.5 mg/dL from baseline within the prior 7 days before RHC
* Chronic kidney disease with eGFR <20 ml/min/1.73 m2
* non-kidney failure requiring extracorporeal or peritoneal ultrafiltration for diuretic-resistant volume overload
* if they had received non-steroidal anti-inflammatory drugs or intravenous contrast within 72 hours before RHC
* prediagnosed glomerulonephritis
* polycystic kidney disease
* postrenal obstruction
* single kidney (functional or anatomical)
* solid organ transplantation
* anticipated life expectancy of <12 months
* likelihood of receiving advanced therapy (mechanical circulatory assist device/lung or cardiac transplant)
* pregnancy or possibility of pregnancy in the next 12 months
* inability to cooperate with respiratory maneuvers during renal Doppler
* refusal to participate
* not available for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients admitted at University Hospital Giessen and Marburg, Campus Giessen with suspected or pre-diagnosed PH undergoing RHC
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse kidney events | Baseline to 12 months
  Number of patients experiencing ≥q of the individual outcomes of the composite outcome of eGFR decline ≥25%, initiation of dialysis, or all-cause mortality

SECONDARY OUTCOMES:
Initiation of dialysis | Baseline to 12 months
  Number of patients requiring initiation of dialysis during follow-up
All-cause mortality | Baseline to 12 months
  Number of patients experiencing all-cause mortality during follow-up
Kidney function decline | 12 months
  Number of patients with eGFR decline ≥25% from baseline

OTHER OUTCOMES:
Worsening PH | Baseline to 12 months
  Number of patients experiencing worsening of PH, defined as hospitalization due to acute right heart failure, increase in PH-targeted medication or diuretics (outpatient or inpatient), worsening of PH as diagnosed by right heart catheterization, or cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Faeq Husain-Syed, MD, Principal Investigator — University of Giessen
Locations (1):
- University Hospital Giessen and Marburg, Campus Giessen, Department of Internal Medicine II, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Husain-Syed F, DiFrancesco MF, Deo R, Barr RG, Scialla JJ, Bluemke DA, Kronmal RA, Lima JAC, Praestgaard A, Tracy RP, Shlipak M, Kawut SM, Kim JS. Associations between eGFR and albuminuria with right ventricular measures: the MESA-Right Ventricle study. Clin Kidney J. 2023 Apr 21;16(9):1508-1520. doi: 10.1093/ckj/sfad096. eCollection 2023 Sep. PMID 37664568
- [Result] Chakinala MM, Coyne DW, Benza RL, Frost AE, McGoon MD, Hartline BK, Frantz RP, Selej M, Zhao C, Mink DR, Farber HW. Impact of declining renal function on outcomes in pulmonary arterial hypertension: A REVEAL registry analysis. J Heart Lung Transplant. 2018 Jun;37(6):696-705. doi: 10.1016/j.healun.2017.10.028. Epub 2017 Nov 6. PMID 29174533